CLINICAL TRIAL: NCT00976807
Title: A Randomised Controlled Trial of Rehabilitation Following Critical Illness: A Short Term Feasibility and Follow-Up Pilot Study
Brief Title: Rehabilitation Following Critical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bronwen Connolly, Clinical Research Fellow, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ1 09/N153
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Critical Illness Myopathy
Keywords: critical care; intensive care; weakness; myopathy; paresis; rehabilitation
MeSH Terms: conditions — Asthenia; Muscular Diseases; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): Pulmonary Rehabilitation
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Eight week programme of twice-weekly (sixteen sessions) supervised exercise and education sessions. Exercise will include aerobic cardiovascular and upper and lower limb strengthening exercises. Each session will comprise a warm-up period, followed by individualised exercises, and completed with a cool-down, and last approximately 40minutes.
  Aerobic exercise will be prescribed based on the results of walking tests and include walking, step-ups, cycling, and strength prescription according to the repetition maximum principle. Patients will complete three sets using this weight.
  Furthermore Borg scores will be used within each session to guide and direct exercise intensity. A home exercise programme will also be designed and accompanied by a manual detailing the individual warm-up, exercises and cool-down, and diary sections to record independent activity.
  Each session will also include an education session where relevant.
  Arms: Intervention

SUMMARY:
The principal research question to be answered by this study is whether an exercise based rehabilitative intervention following critical illness can generate improvements in exercise capacity and quality of life beyond current (usual) care. The investigators will also aim to demonstrate that such an intervention is both practical and cost-effective.

DETAILED DESCRIPTION:
Advances in medicine mean that an increasing number of critically ill people, including those with severe pneumonia (lung infection), chronic obstructive pulmonary disease (also known as emphysema or chronic bronchitis) or the "acute respiratory distress syndrome", survive admission to the hospital intensive care unit. Survivors report health problems such as breathlessness and weakness long after discharge. In a study monitoring over 800 patients discharged from an intensive care ward, over half required some form of caregiver assistance after 1-year.

Whilst on intensive care, patients usually require help to breathe from a ventilator machine and become immobilised. This leads to weak breathing muscles in three quarters of patients, as well as weak and wasted arm and leg muscles. Survivors struggle to regain their previous level of daily activity and function, limited by shortness of breath, muscle weakness and tiredness. It is recognised that people with chronic lung problems, such as chronic obstructive pulmonary disease, face similar problems. In this condition, exercise based therapy has been shown to improve muscle strength, walking ability, shortness of breath, and importantly quality of life.

Given these experiences, a new trial will evaluate a novel programme of exercise-based rehabilitation training in patients discharged from intensive care. The programme will last for 8-weeks and will use exercises designed to correct the breathing and limb muscle weakness, as well as education to help patients cope more effectively. The programme will begin as soon as possible following discharge from hospital and will be conducted on a mostly outpatient basis until the course is completed. By speeding the recovery of strength and activity, it is anticipated that quality of life will be improved, which this trial will attempt to measure.

The rehabilitation programme will include aerobic cardiovascular, and upper and lower limb strengthening exercises, in addition to relevant education sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years AND admitted to critical care unit
* Ventilated >48-hours (via endotracheal tube) OR received continuous non- invasive ventilation (NIV)/non-invasive continuous positive airways pressure (CPAP)
* Admitted to ICU > 48-hours and evidence of SIRS
* Glasgow Coma Score (GCS) 15 (of 15) AND Abbreviated Mini-Mental Test Score (AMMTS) >/= 8 (of 10) on enrolment into rehabilitation programme
* Mobilising on ward to a degree sufficient as to begin a majority of proposed exercises. Clinical stability for observed exercise as judged by trial team is a prerequisite.
* Participant willingness to complete a programme of exercise based therapy aimed at reducing weakness and shortness of breath: subjective weakness or dyspnoea relative to their pre-admission state is implicit

Exclusion Criteria:

* Patients referred for terminal care or prognosis likely to be less than 12-months
* Unstable coronary artery syndrome
* Limb amputation (given special requirement for orthotics/rehabilitation)
* Critical peripheral vascular disease awaiting re-vascularisation procedure (or claudication distance <100 metres)
* Stroke with hemiparesis (likely need for specialised rehabilitation/stay on stroke unit)
* Severe, disabling locomotor problem or severe burns, which prevent effective participation in the exercises contained in the rehabilitation programme.
* Psychiatric disease necessitating anti-psychotic medication, deliberate drug overdose as the admitting ICU indication, ongoing treatment for drug or alcohol addiction, persons of no fixed abode post-discharge
* Patients undergoing renal haemodialysis (given the associated commitment to outpatient attendance)
* Extra contractual ICU referral (only if distance greater than suitable for twice weekly travel)

Additional exclusion criteria for muscle biopsy samples:

* Coagulopathy e.g. warfarin use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incremental Shuttle Walk Test | Eight weeks

SECONDARY OUTCOMES:
Health Related Quality of Life | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, BSc (Hons), MBBS, MRCP, PhD, Study Director — St.Thomas' Hospital
Locations (2):
- United Kingdom (2):
  - St.Thomas' Hospital, London, London
  - King's College Hospital, London, London

REFERENCES:
- [Derived] Connolly B, Thompson A, Douiri A, Moxham J, Hart N. Exercise-based rehabilitation after hospital discharge for survivors of critical illness with intensive care unit-acquired weakness: A pilot feasibility trial. J Crit Care. 2015 Jun;30(3):589-98. doi: 10.1016/j.jcrc.2015.02.002. Epub 2015 Feb 7. PMID 25703957